CLINICAL TRIAL: NCT06220383
Title: Evaluation of The Effect of Crowns Applied wıth Hall Technique on Occlusion: Randomized Clinical Study
Brief Title: Evaluation of The Effect of Crowns Applied With Hall Technique on Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Funda Cagırır Dindaroglu, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-TDU-DİŞF-0013
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Child, Only; Quality of Life
Keywords: Hall technique; Paediatric dentistry; Stainless Steel

STUDY DESIGN:
Intervention Model Description: Randomized controlled, double-blind clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was performed by a computer-generated random sorting sequence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall technique (Experimental): In the Hall technique method, an orthodontic separator was placed 2 days before the procedure to create distance for the crown in the mesial and distal contact areas of the tooth on which the crown will be placed. A stainless steel crown was cemented on the tooth with glass ionomer cement without local anesthesia, caries cleaning or any preparation. The participant was asked to close the teeth tightly for 2-3 minutes.
  Interventions: Procedure: Hall technique
- Conventional technique (Active Comparator): In the conventional technique, after the area to be anesthetized was dried, topical anesthetic solution (Locanest 10% spray lidocaine, Avixa, Turkey) was applied to the mucosa with a cotton pellet for one minute. For infiltrative anesthesia, 4% articaine solution (Ultracaine DS Forte ampoule, Sanofi-Aventis GmbH, Germany) containing 1 ml of 1:100,000 epinephrine was applied. Preparation was made on the mesial, distal and occlusal sides of the tooth. The decay was cleaned and the cavity was filled with glass ionomer cement (Ketac Molar Easymix, 3M™ ESPE™, St. Paul, MN, USA). The stainless steel crown was bonded with glass ionomer cement (Ketac Cem Easymix, 3M™ ESPE™, St. Paul, MN, USA).
  Interventions: Procedure: Conventional technique

INTERVENTIONS:
Procedure: Hall technique — Prepless crown technique
  Arms: Hall technique
Procedure: Conventional technique — 1 or 1,5 mm preparation on mesial, distal and occlusal of the tooth
  Arms: Conventional technique

SUMMARY:
This study aims to evaluate and compare the change on occlusion after placing stainless steel crowns (SCC) using Hall technique and conventional technique in children between the ages of 5-8. In addition, the investigators planned to analyze the change in oral health-related quality of life between SCC applied with the Hall technique and SCC applied with the conventional method, before and after clinical application.

DETAILED DESCRIPTION:
First, the participants who met the inclusion criteria were included in 2 study groups according to age, gender, dental experience, tooth number, applied stainless steel crown technique, Decayed, Missing due to caries, and Filled teeth in the permanent teeth/decayed, missing due to caries, and filled teeth in the deciduous teeth (DMFT/dmft index) values and International Caries Detection and Assessment System (ICDAS II) and radiographic evaluation criteria. In the experimental group, stainless steel crowns were placed on the teeth of 39 participants using the Hall technique. In the control group, stainless steel crowns were placed on the teeth of 39 participants using conventional technique.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with American Society of Anesthesiologists score I (ASA I),
* Subjects with Frankl's behavior rate III (positive) and IV (definitely positive),
* Clinically, Black class II enamel-dentin caries in the upper jaw primary second molar is; ICDAS II Scale score 4, score 5 and the accepted values in the evaluation of radiographic dental caries are D1-RA3, D2-RB4, D3-RC5,
* Antagonist of the tooth planned to be processed,
* Lamina dura and periodontal space can be observed normally
* There is permanent tooth germ underneath or the position is normal.

Exclusion Criteria:

* Allergic to the local anesthetics or sulfites,
* Had teeth with pain or sepsis,
* Were uncooperative during clinical examination,
* TMJ disorder,
* Had parafunctional habit

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
The measurement of intrusion of teeth with stainless steel crown applied with Hall technique using Gom Inspect | Immediately before the procedure and one month control
  Intrusion scores in Hall technique 0-3, where 0 means no movement, 3 means intrusion
The measurement of intrusion of teeth with stainless steel crown applied with conventional technique using Gom Inspect | Immediately before the procedure and one month control
  0-3, where 0 means no movement, 3 means extrusion
Change from measurement the distance between the cusps of canines with stainless steel crown applied with Hall technique using Exocad | Immediately before the procedure and one month control
  0-2, where 0 means no movement, 2 means no closure
Change from measurement the distance between the cusps of canines with stainless steel crown applied with conventional technique using Exocad | Immediately before the procedure and one month control
  0-2, where 0 means no movement, 2 means no closure

SECONDARY OUTCOMES:
Measuring the impact of stainless steel crowns on oral health and quality of life in children section with the Early Childhood Oral Health Impact Scale | Immediately after the procedure and one month control
  Child sections have a possible range from 0 to 36. 0=Never or hardly ever 36= Occasionally, often, or very often
Measuring the impact of stainless steel crowns on oral health and quality of life in parents section with the Early Childhood Oral Health Impact Scale | Immediately after the procedure and one month control
  Family sections have a possible range from 0 to 16. 0=Never or hardly ever 16= Occasionally, often, or very often

CONTACTS AND LOCATIONS:
Locations (1):
- Funda Çağırır Dindaroğlu, Izmir, Turkey (Türkiye)